CLINICAL TRIAL: NCT02682251
Title: Engaging Patients in Heart Failure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Health (Other)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Principal Investigator, Tammy Toscos, Research Scientist, Informatics, Parkview Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRC15-0904 BTK
Record Dates: First submitted 2016-01-27; First posted 2016-02-15 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Congestive Heart Failure
Keywords: Cardiac Resynchronization Therapy Devices; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart Failure Patients with CRT-CIED (Experimental): PHR Messaging to notify patient of device transmitted information (i.e. percentage LV pacing)
  Interventions: Other: PHR Messaging

INTERVENTIONS:
Other: PHR Messaging — PHR messaging of data pertinent to chronic resynchronization therapy and heart failure management (i.e. percentage LV pacing).

SUMMARY:
An interventional study to empower congestive heart failure patients who have a cardiac resynchronization therapy-cardiac implantable electronic device (CRT-CIED) by using a personal health record (PHR) to directly message them their device data and send alerts based on percent left ventricular pacing.

DETAILED DESCRIPTION:
An interventional study to empower congestive heart failure patients who have a cardiac resynchronization therapy-cardiac implantable electronic device (CRT-CIED) by using a personal health record (PHR) to directly message them their device data and send alerts based on percent left ventricular pacing.

There will be three phases in this study. In the first phase the investigators will employ a user-centered design approach to better understand what types of information that patients who have a remotely monitored CRT-CIED would find beneficial towards understanding and managing their disease. The investigators also hope to uncover expectations for alert mechanisms and two-way messaging between provider and patient around CIED remote monitoring data. In the second phase the investigators will implement the PHR intervention as designed in phase 1. In the third phase of this study, the investigators will test the PHR intervention in a single arm, 6-month trial.

A maximum of 120 participants (including patients and their caregiver, partner, and/or support persons) will be enrolled in the focus groups for phase 1. A maximum of 10 patients will be enrolled in the design session to follow in phase 1. After building the intervention in phase 2, a maximum of 30 patients will be enrolled in the technology trial for phase 3. Enrollment is projected to be complete within six months for phase 1, and within one year for phase 3.

In phase 3, adult subjects (N=30) with a diagnosis of congestive heart failure undergoing chronic resynchronization therapy through their CIED will receive interventional messaging through their PHR regarding percent left ventricular pacing.

The study duration will commence at the time of informed consent documentation during the first focus group and conclude at the time of the last patient visit during the technology trial.

Impact of PHR messaging will be evaluated by timeliness of patient calls to clinic for adjustment in therapy, an improved percentage of LV pacing over 6 months compared to historical controls from the same clinic, as well as self-reported patient engagement. Timeliness of patient calls to clinic will be evaluated through record of patient calls to clinic 6 months prior to study and 6 months during study. Patient engagement will be evaluated through patient survey at start and end of study.

Patients will follow standard of care + intervention during study.

ELIGIBILITY:
FOCUS GROUPS

Inclusion Criteria:

1. Remotely monitored with CRT-CIED

   * focus groups 1 & 2: implant ≤ 12 months
   * focus groups 3 & 4: implant ≥ 12 months
2. Current patient of PPG-Cardiology
3. History of HFrEF (heart failure in the setting of reduced ejection fraction)
4. Access to computer and internet
5. *Ability to provide informed consent
6. *Age ≥ 18 years

   * 5 and 6 must apply to caregivers, partners, and/or support persons

Exclusion Criteria:

1. Not remotely monitored with CRT-CIED
2. Not current patient of PPG-Cardiology
3. No history of HFrEF
4. Pacemaker dependent
5. Does not have access to computer and internet
6. *Inability to provide informed consent
7. *Age < 18 years
8. *Does not meet inclusion criteria

   * Only 6, 7, and 8 apply to caregivers, partners, and/or support persons

TECHNOLOGY TRIAL

Inclusion Criteria:

1. Remotely monitored with Biotronik CRT-CIED for more than 60 days
2. Ability to provide informed consent
3. Age ≥ 18 years
4. Willing to have MyChart or proxy to MyChart
5. Current patient of PPG-Cardiology
6. History of HFrEF

Exclusion Criteria:

1. Do not have a Biotronik CRT
2. Have a Biotronik CRT-CIED for less than 60 days
3. Not being remotely monitored with a Biotronik CRT-CIED
4. No history of HFrEF
5. Inability to provide informed consent
6. Age < 18 years
7. Lack of internet access or otherwise unable to access MyChart
8. Pacemaker dependency
9. Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Timeliness of calls to clinic for adjustment in therapy | 6 months during study
Patient engagement evaluated through patient survey | 6 months during study
Improved percentage of LV pacing | 6 months during study

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Toscos, PhD, Principal Investigator — Parkview Health; Michael Mirro, MD, Principal Investigator — Parkview Health
Locations (1):
- Parkview Health, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.